CLINICAL TRIAL: NCT06439004
Title: The Use of Quantitative Sensory Testing to Characterize Somatosensory Functionality
Brief Title: The Use of QST to Characterize Somatosensory Functionality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S69194
Record Dates: First submitted 2024-05-27; First posted 2024-06-03 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy volunteers (Experimental): Healthy volunteers to evaluate the inter-period reproducibility of thirteen QST parameters.
  Interventions: Other: Quantitative Sensory Testing

INTERVENTIONS:
Other: Quantitative Sensory Testing — Performing QST on the dominant hand, right forearm, right flank and lower back.

SUMMARY:
Pain has a significant impact on quality of life and poses an enormous burden on the healthcare system. The subjective nature of pain complicates its mapping and treatment. Quantitative Sensory Testing (QST) aims to characterize the somatosensory phenotype using calibrated stimuli and subjective thresholds. This set of procedures enables quantification of the somatosensory function in small fibers (thinly myelinated Aδ and unmyelinated C), as well as large fibers (thickly myelinated Aβ). In this way, sensory loss (hypoesthesia, hypoalgesia) or sensory gain (hyperesthesia, hyperalgesia, allodynia) can be detected.

In this study, the inter-period reproducibility of thirteen QST parameters will be determined on the dominant hand, right forearm, right flank and lower back of 20 healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent has been obtained prior to any screening procedures.
* Subject is ≥ 18 years and ≤ 25 years of age.
* Subject is a non-smoker for at least 6 months before the start of the study.
* Subject has a body mass index (BMI) between 18-30 kg/m².
* Subject is in good general health, based on medical history and vital signs.

Exclusion Criteria:

* Subject has a history of any illness which, in the investigator's opinion, might confound the results of the study, including conditions which affect the normal somatosensory functionality.
* Subject has eczema, scleroderma, psoriasis, dermatitis, or any other abnormality on the skin of the dominant hand, right forearm, right flank or lower back which, in the investigator's opinion, might interfere with the study assessments.
* Subject is unable to refrain from drinking alcohol 24 hours prior to each study visit, is currently a user of drugs, or has a history of alcohol and/or drug abuse.
* Subject is unable to refrain from drinking caffeinated beverages 24 hours prior to each study visit.
* Subject has used concomitant drugs and/or treatments that may interfere, in the investigator's opinion, with the study results.
* Subject is in a situation or has a condition which, in the investigator's opinion, may interfere with safe and optimal participation in the study.
* Female subject who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and is not using an adequate contraceptive method.
* Subject is participating in another trial which, in the investigator's opinion, might confound the results of the study.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-09-12 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Inter-period reproducibility of QST | Interval of 7 - 21 days between both periods
  Inter-period reproducibility of thirteen different QST parameters on the dominant hand, right forearm, right flank and lower back of healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Jan de Hoon, MD, PhD, MSc, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No